CLINICAL TRIAL: NCT03350516
Title: Demonstrating Non-inferiority of Lower Dose Calcium Supplementation During Pregnancy for Reducing Preeclampsia and Neonatal Outcomes
Brief Title: Non-inferiority of Lower Dose Calcium Supplementation During Pregnancy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: St. John's Research Institute (Other); Ifakara Health Institute (Other); Africa Academy for Public Health (Other)
Responsible Party: Principal Investigator, Wafaie Fawzi, Richard Saltonstall Professor of Population Sciences, Professor of Nutrition, Epidemiology, and Global Health, Chair of the Department of Global Health and Population, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: OPP1172660
Record Dates: First submitted 2017-11-19; First posted 2017-11-22 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Pregnancy Related
MeSH Terms: interventions — Calcium; Calcium Carbonate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Daily 500 mg Calcium (Experimental)
  Interventions: Dietary Supplement: Daily 500 mg elemental calcium as calcium carbonate
- Daily1500 mg Calcium (Standard dose) (Active Comparator)
  Interventions: Dietary Supplement: Daily1500 mg elemental calcium as calcium carbonate

INTERVENTIONS:
Dietary Supplement: Daily 500 mg elemental calcium as calcium carbonate — Pregnant women in this arm will be provided and counselled to take three tablets, one containing 500 mg elemental calcium as calcium carbonate and 2 placebo supplements daily (total of 500 mg daily). The supplements in India will also contain 83.3 IU each of vitamin D3, for a total of 250 IU daily. No vitamin D3 will be given in Tanzania.
  Arms: Daily 500 mg Calcium
Dietary Supplement: Daily1500 mg elemental calcium as calcium carbonate — Pregnant women in this arm will be provided and counselled to take three tablets each containing 500 mg elemental calcium as calcium carbonate daily (total of 1500 mg daily) as currently recommended by the World Health Organization. The supplements in India will also contain 83.3 IU each of vitamin D3, for a total of 250 IU daily. No vitamin D3 will be given in Tanzania.
  Arms: Daily1500 mg Calcium (Standard dose)

SUMMARY:
The World Health Organization currently recommends that pregnant women in populations with low calcium intake receive daily calcium supplementation (1500 - 2000 mg) divided into three doses which are preferably taken at mealtimes, in addition to daily iron folic-acid supplements. Despite proven efficacy and the WHO recommendation, calcium supplementation in pregnancy is not standard of care in the vast majority of low-income and middle-income countries. Two important barriers to implementation are the cost of the supplements and complexity of the suggested calcium dosing schedule. A lower dose of calcium (500 mg) administered as a single dose has been shown to be beneficial in several trials, and if found to be as effective as the 1500 mg supplementation regimen, it may help overcome these barriers and increase individual and health system adoption.

The Investigators will conduct two parallel, individually randomized, double blind non-inferiority trials in India and Tanzania. Participating pregnant woman will be randomized to either 1500 mg or 500 mg calcium supplementation. The India and Tanzania trials are independently powered for the primary outcomes of i) preeclampsia and ii) preterm birth. The India and Tanzania sites will each enroll 11,000 participants.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous
* Attending first ANC visit at study clinics
* Pregnant women <20 weeks
* ≥ 18 years old
* Intending to stay in study area until 6 weeks post delivery
* Provides informed consent

Exclusion Criteria:

* History or signs and/or symptoms of nephrolithiasis
* Prior diagnosis of parathyroid disorder or thyroidectomy
* Diseases that require digoxin, phenytoin, or tetracycline therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22000 (Actual)
Dates: Start 2018-11-30 (Actual); Primary Completion 2022-11-03 (Actual); Study Completion 2022-12-16 (Actual)

PRIMARY OUTCOMES:
Proportion of pregnant women with incident preeclampsia | Gestational week 20 to Delivery
Proportion of preterm birth | Birth

CONTACTS AND LOCATIONS:
Overall Officials: Wafaie W Fawzi, MBBS, DrPH, Principal Investigator — Harvard School of Public Health (HSPH)
Locations (3):
- St. John's Research Institute, Bangalore, India
- Tanzania (2):
  - Africa Academy for Public Health, Dar es Salaam
  - Ifakara Health Institute, Dar es Salaam

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Dwarkanath P, Muhihi A, Sudfeld CR, Wylie BJ, Wang M, Perumal N, Thomas T, Kinyogoli SM, Bakari M, Fernandez R, Raj JM, Swai NO, Buggi N, Shobha R, Sando MM, Duggan CP, Masanja HM, Kurpad AV, Pembe AB, Fawzi WW. Two Randomized Trials of Low-Dose Calcium Supplementation in Pregnancy. N Engl J Med. 2024 Jan 11;390(2):143-153. doi: 10.1056/NEJMoa2307212. PMID 38197817
- [Derived] Pembe AB, Dwarkanath P, Kikula A, Raj JM, Perumal N, Paulo HA, M R, Duggan CP, Masanja HM, Chopra N, Sando MM, Thomas T, Yelverton CA, Muhihi A, Kurpad AV, Fawzi WW, Wylie BJ, Sudfeld CR. Hypertensive disorders of pregnancy and perinatal outcomes: two prospective cohort studies of nulliparous women in India and Tanzania. BMJ Glob Health. 2025 Jul 10;10(7):e016339. doi: 10.1136/bmjgh-2024-016339. PMID 40639854
- [Derived] Dwarkanath P, Muhihi A, Sudfeld CR, Rani S, Duggan CP, Sando MM, Wylie BJ, Fernandez R, Kinyogoli S, Munk C, Perumal N, Raj JM, Buggi N, Swai N, Thomas T, Wang M, Kurpad AV, Masanja H, Pembe AB, Fawzi WW. Non-inferiority of low-dose compared to standard high-dose calcium supplementation in pregnancy: study protocol for two randomized, parallel group, non-inferiority trials in India and Tanzania. Trials. 2021 Nov 24;22(1):838. doi: 10.1186/s13063-021-05811-7. PMID 34819147